CLINICAL TRIAL: NCT06972550
Title: Volar Locked Plating for Distal Radius Fractures: Should the Pronator Quadratus Be Spared?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-837-2018
Record Dates: First submitted 2025-05-03; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pronator Quadratus sparing (Experimental): The pronator quadratus was spared during ORIF of the fracture
  Interventions: Procedure: pronator quadratus sparing

INTERVENTIONS:
Procedure: pronator quadratus sparing — the pronator quadratus was spared when doing orif and the plare was slided beneath it

SUMMARY:
Volar locked plates for the distal radius fractures (DRFs) are applied through the Henry approach and it's modification, this approach entails a routine step to disinsert the pronator quadratus from it's radial and distal attachment. This muscle insertion is mostly fleshy with minimal tendinous tissue and surgeons find it difficult to reattach at the end of the surgery, the hardware come in direct contact with the flexor tendons.

DETAILED DESCRIPTION:
Distal radius fractures (DRFs) account for about 17.5% of all adult fractures and represent the most common fracture of the upper extremity. For severely displaced or unstable fractures, open reduction and internal fixation (ORIF) is often indicated. Volar locking plate fixation through the flexor carpi radialis (FCR) approach is widely used and considered a standard technique for distal radius fixation. Classically, the pronator quadratus (PQ) muscle is released from the radial side of the distal radius to expose the fracture and is later repaired after plate fixation. However, this repair is often not feasible or reliable. Some authors have suggested that failure to restore the PQ may leave the plate exposed to the flexor tendons, increasing the risk of tendon irritation or rupture.

To address these concerns, minimally invasive PQ-sparing approaches have been developed. Imatani et al. first described a technique for volar plating without detaching the PQ, and Dos Remedios et al. reported a similar approach. Theoretically, preserving the PQ creates a cushion between the plate and the flexor tendons and maintains the muscle's function. Several studies have reported better early functional outcomes and less pain post-operatively with PQ-sparing than the traditional approach.

In this prospective case series at a Level I trauma center with a dedicated hand surgery service, the PQ-sparing volar plating technique for distal radius fractures is evaluated. The study's main objectives were to determine whether the PQ can be preserved without compromising fracture reduction, to describe how a volar locking plate can be applied without releasing the PQ, to identify potential benefits of PQ preservation, and to assess any drawbacks of this approach.

ELIGIBILITY:
Inclusion Criteria:

* isolated closed distal radius fractures

Exclusion Criteria:

* fractures >3 weeks old,
* age >60 years (reflecting our practice of treating most low-demand elderly patients nonoperatively unless the fracture was highly unstable),
* pathologic fractures (e.g. metastatic lesions).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Radiological bone union | 2 months, 4 months
  an xray was done to determine if the bone ends had become united.

SECONDARY OUTCOMES:
pain postoperatively by the Visual Analogue Scale (VAS) score | 2 months, 4 months
  pain is measured by a vas score both post operative and throughout the follow up period in a 10 point scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes